CLINICAL TRIAL: NCT03744650
Title: Improving Awareness, Knowledge and Heart-related Lifestyle of Coronary Heart Disease Among Working Population Through a mHealth Programme
Brief Title: mHealth Lifestyle Intervention on CHD Primary Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Wang Wenru, A/Prof, National University of Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-15-059
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: CHD - Coronary Heart Disease; Health Knowledge, Attitudes, Practice; Health Behavior
Keywords: Pirmary prevention; Coronary Heart Disease; mHealth
MeSH Terms: conditions — Coronary Artery Disease; Behavior; Health Behavior; Coronary Disease

STUDY DESIGN:
Intervention Model Description: A two-phase study design will be adopted. Phase 1 is a pilot, two-arm randomized controlled trial (RCT) study and phase 2 is a single group pretest and repeated posttest longitudinal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Care4Heart" programme (Experimental): The single group pretest and repeated posttest longitudinal study design is adopted in the main study. All the recruited participants received the study intervention
  Interventions: Behavioral: "Care4Heart" programme

INTERVENTIONS:
Behavioral: "Care4Heart" programme — A 4-week mHealth programme in the form of a smartphone app, named "Care4Heart", has been developed. The content and scope of the design are developed by a thorough literature review and an extensive analysis of existing education leaflets and brochures used to prevent CHD. The contents are specified and tailored to the working population.
  The app is developed by a team of software engineers from Computing School of NUS. Several functions include: (1) app using instructional video; (2) easy-to-read information on healthy lifestyle toward heart health, including information about the disease, CHD risk factors (e.g. diet, smoking cessation), stress, physical exercises and relaxation techniques; and (3) scheduled reminders for doing exercise and relaxation

SUMMARY:
Background: Coronary heart disease (CHD), the most prevalent type of cardiovascular disease among adults, has been identified as one of the chronic diseases which are epidemic in the world. Teaching and encouraging the working population to adopt a healthier lifestyle could favor in preventing and/or decreasing the incidence of CHD among this population. The use of mobile application (app) is the next logical wave of healthcare support tools to prevent and manage chronic diseases like CHD.

Aims: The aims of the study are to develop a mHealth programme, entitled "Care4Heart" for the working population in Singapore, and thereafter examine its feasibility and effectiveness in increasing the awareness and knowledge of coronary heart disease (CHD) as well as improving their heart-related lifestyle.

Methods: A two-phase study design will be adopted. Phase 1 is a pilot, two-arm randomized controlled trial (RCT) study and phase 2 is a single group pretest and repeated posttest longitudinal study. The study will be conducted in National University of Singapore. A convenience sampling will be used, and a total of 240 healthy working adults will be recruited via posters advertising in campus canteens, which comprising 80 participants in Phase 1 and 160 participants in Phase 2 study. The first recruited 80 participants will be randomly allocated to an intervention group and a control group, and only those in the intervention group will receive 4-week "Care4Heart" programme. For the participants recruited in phase 2 (n = 160), the newly developed mobile app will be installed onto their' smartphones, and a well-trained research assistant will brief the participants about the utilization of the app.

The main outcomes will be measured using the survey questionnaires: Awareness of CHD, Heart Disease Fact Questionnaire-2, Behavioral Risk Factor Surveillance System and Perceived Stress Scale. Data will be collected at baseline, and at the 4th week for phase 1 study while a third data collection at the 6th month thereafter will be conducted for phase 2 participants. Data will be analyzed using IBM SPSS 22.0.

Applications: If this project is proved to be feasible and effective, "Care4Heart" app, a novel CHD prevention programme will be popularized nationwide to promote knowledge and elicit positive heart-related behavioral changes for the working population in Singapore

DETAILED DESCRIPTION:
The study aims to develop a mHealth programme, entitled "Care4Heart" for the working population in Singapore and examine its feasibility and effectiveness in increasing the awareness and knowledge of coronary heart disease (CHD) as well as improving their heart-related lifestyle.

The objectives are:

1. To develop a mHealth programme using the smartphone app, entitled "Care4Heart" for the working population in Singapore to assist them in establishing a healthy lifestyle.
2. To test the effectiveness of the "Care4Heart" app in increasing the awareness and knowledge of CHD among the working population in Singapore.
3. To test the effectiveness of the "Care4Heart" app in eliciting a positive heart-related lifestyle modification, including stress reduction among the working population in Singapore.

Background Deaths caused by CHD are often preventable. Deranged serum lipid profile, hypertension, obesity, physical inactivity and excess working stress are the well-known preventable risk factors of CHD, and the reduction of these risk factors will improve physical and psychological health and prevent future adverse and fatal cardiac events. Sedentary lifestyles and unhealthy diets are common reasons that may predispose Singaporeans to the risk of developing CHD, especially the majority of the workforce working in offices who engage in little or no physical activity. It was reported that about 40% of the working population (i.e. 21 to 65 years old) in Singapore do not engage in regular physical exercise. The increasing popularity of high fat diet and eating out and the high levels of stress experienced by the working population may further increase their risk of developing CHD.

Many of risk factors of CHD are modifiable and can be greatly reduced by adopting a healthy lifestyle. Exercising regularly and following a healthy diet plan are effective strategies in lowering cardiovascular risk factors. Obviously there is a need for an updated educational programme aimed at teaching and encouraging people in the working population to adopt a healthier lifestyle, which would result in them changing their behaviours and sustaining a healthy lifestyle to reach optimal health. Even though, health promotion programmes including the traditional face-to-face cardiac education sessions have been developed to be accessed by the general population, a known barrier for not reaching the working population is the lack of time as a result of long work hours. With a substantial increase in the number of people owning smartphones and a sharp increase in the usage of smartphones in recent years, the smartphone is a device most people in Singapore own. Recently the Infocomm Development Authority of Singapore (2013) announced plans for a well-connected mobile network to support major industries including healthcare. Hence the promotion of mobile health (mHealth) is the next logical wave of healthcare support tools to prevent and manage chronic diseases like CHD. A recent whitepaper based on market research conducted in Singapore reported that about 92% of Singaporeans aged between 25 to 39 years owned smartphones. While 83% of the older population aged from 55 years onwards owned smartphones as well. Based on this report, it is widely expected that mHealth will reach many Singaporeans as tools to maintain and improve their health.

Over the past few decades, more innovative ways for the design and delivery of primary/secondary prevention programme have been developed due to the rapid evolution of technology. One such programme used increasingly in the prevention and management of chronic diseases is mHealth which includes web-based programmes and smartphone applications (apps). Several studies conducted in Western countries reported on the effectiveness of mHealth in improving self-management skills and increasing healthy behaviours of individuals with chronic disease, such as diabetes, hypertensionand CHD. More importantly, apps are more accessible and convenient, enabling the information to reach more people by overcoming obstacles such as physical distance to attend a face-to face education session. However, these apps that have been developed are not completely relevant and suitable for Singaporeans because of significant cultural and economic differences that influence cardiac risk factors. For example the diet in Singapore and the culture of longer working hours are significantly different from Western countries.

Design/Methodology This study was funded by a grant from Singapore Heart Foundation (Grant Number: RG2013/02). A two-phase study design will be adopted. Phase 1 is a pilot, two-arm RCT study and phase 2 is a single group repeated test longitudinal study. The data of Phase1 study will be collected at the baseline and 4th week. The Phase 2 data will be collected at the baseline, 4th week and 6th months from the baseline.

Participants

The target population for this study is the working population in Singapore. The study will be conducted in National University of Singapore. A total of 240 convenient samples will be recruited via posters advertising in campus canteens, comprising 80 subjects in Phase 1 and 160 subjects in Phase 2 study. The first recruited 80 participants will be randomly allocated to an intervention group or a control group.

Phase 1 Randomization All eligible participants will be assigned a unique case number according to the sequence in which participants are recruited, for example, the first eligible participant will be assigned the number of one, and the second eligible assigned the number of two and so on. A total of 40 numbers without any duplicates will be randomly generated, from 1 to 80, using SPSS. Participants whose assigned numbers matched the numbers generated by the software will be allocated into the intervention group; otherwise, the participant will be assigned to the control group.

Theoretical rationale for intervention According to the Health Belief Model, there are several factors which influence health outcomes of an individual. These factors are: (1) the individual's belief that there is a threat to his/her health because of the illness, (2) the level of motivation of the individual to take action to improve his/her health and (3) the individual's belief that the intervention recommended will decrease the threat to his/her health. These factors will be addressed in our proposed "Care4Heart" mHealth programme which will cover the CHD risk factors, the possible health-threatening outcomes and strategies to decrease these risk factors are provided.

Intervention A 4-week mHealth programme in the form of a smartphone app, named "Care4Heart", has been developed. The content and scope of the design are developed by a thorough literature review and an extensive analysis of existing education leaflets and brochures used to prevent CHD. The contents are specified and tailored to the working population.

The app is developed by a team of software engineers from Computing School of NUS. Several functions include: (1) app using instructional video; (2) easy-to-read information on healthy lifestyle toward heart health, including information about the disease, CHD risk factors (e.g. diet, smoking cessation), stress, physical exercises and relaxation techniques; and (3) scheduled reminders for doing exercise and relaxation.

A website (www.care4heart.sg) has been created as well. Participants are allowed to visit the website for the details about this project and research team members.

Study procedure

Phase 1: Pilot RCT One face-to-face briefing session will be offered for the 40 participants allocated to the intervention group after the consent is obtained. The smartphone app will be installed to the participant's own smartphone, and one of the research team members will brief the participant on the utilization of app. This session will take about 20 to 30 minutes. After participants are familiar with the setup and the structure of the app, the participants will be expected to spend 15-20 minutes every day to go through all the educational content in 4 weeks' time. The participants will also be encouraged to change their lifestyle to modify their cardiac risk factors according to the information given in the app, for example engaging in regular exercise, and practicing relaxation.

No intervention will be provided to the participants in the control group. Data will be collected online. Participants can complete the questionnaires on the website (www.care4heart.sg). All data will be electronically stored in an encrypted and password accessed-only computer database, in accordance to the University's Research Data Management Policy.

The above questionnaires will be completed at two time points; (1) upon giving consent to participate in the study (baseline), and (2) at the 4th week.

Phase 2: single group pretest and repeated posttest longitudinal study A total of 160 participants will be recruited for phase 2 study. The same as phase 1 study, One face-to-face briefing session will be offered for all participants after the consent is obtained. The smartphone app will be installed to the participant's own smartphone, and one of the research team members will brief the participant on the utilization of app. This session will take about 20 to 30 minutes. . After participants are familiar with the setup and the structure of the app, the participants will be expected to spend 15-20 minutes every day to go through all the educational content in 4 weeks' time. The participants will also be encouraged to change the lifestyle to modify their cardiac risk factors according to the information given in the app, for example engaging in regular exercise, and practicing relaxation.

Data will be collected online. Participants can complete the questionnaires on the website (www.care4heart.sg). All data will be electronically stored in an encrypted and password accessed-only computer database, in accordance to the University's Research Data Management Policy.

The above questionnaires will be completed at three time points; (1) upon giving consent to participate in the study (baseline); (2) at the 4th week from the baseline; and. (3) at the 6th month follow-up period.

Data analysis All data obtained will be analyzed using IBM SPSS 22.0 (Armonk, NY, USA). Descriptive statistics, including the frequency distribution, mean and standard deviation will be used to describe the social-demographic and anthropometric data, HDFQ-2, BRFSS and PSS-10 of all participants. In Phase 1 study, significant differences in the change scores of HDFQ-2, BRFSS and PSS-10 will be examined via paired samples t-test and between-group changes will be examined via independent t-test. In Phase 2 study, significant differences in the change scores of HDFQ-2, BRFSS and PSS-10 will be examined via paired samples t-test. The level of significance selected for this study is set at p = 0.05, indicating a 5% of committing a Type I error. The Bonferroni posthoc test will be run to reduce the likelihood of identifying the difference by chance.

ELIGIBILITY:
Inclusion Criteria:

1. working full-time;
2. aged between 21-65 years;
3. use a smartphone (e.g. Samsung, iPhone) in their daily lives frequently; and
4. able to read, speak and understand English.

Exclusion Criteria

1. have a clinical diagnosis of CHD or other heart diseases (e.g. congestive heart failure);
2. work in a health-relevant school/department/environment (e.g. school of medicine, school of public health, department of dentistry, school of pharmacy; university health centre); and
3. have reading difficulties.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Awareness of Coronary Heart Disease | baseline
  Questions that assess participants' awareness of CHD in Singapore will be developed based on the statistic facts of CHD in Singapore, for example: (1) the percentage of deaths by CHD in Singapore; and (2) the second leading cause of death in Singapore
Awareness of Coronary Heart Disease | 4th week from the baseline
  Questions that assess participants' awareness of CHD in Singapore will be developed based on the statistic facts of CHD in Singapore, for example: (1) the percentage of deaths by CHD in Singapore; and (2) the second leading cause of death in Singapore
Awareness of Coronary Heart Disease | 6th months from the baseline
  Questions that assess participants' awareness of CHD in Singapore will be developed based on the statistic facts of CHD in Singapore, for example: (1) the percentage of deaths by CHD in Singapore; and (2) the second leading cause of death in Singapore

SECONDARY OUTCOMES:
Heart Disease Fact Questionnaire-2 (HDFQ-2) | baseline
  Heart Disease Fact Questionnaire-2 (HDFQ-2) is a 25-item measure contains true/false questions that were developed to assess participants' knowledge of major risk factors for the development of CHD. Each true/false question that was correctly answered was scored as 4 points, for a maximum possible score of 100, indicting a higher level of knowledge. Any questions that were either unanswered or unsure were scored as incorrect. The HDFQ-2 has demonstrated adequate internal consistency with Cronbach alpha of 0.84 and good test-rested reliability with intraclass correlation coefficient (ICC) of 0.89.
Heart Disease Fact Questionnaire-2 (HDFQ-2) | 4th week from the baseline
  Heart Disease Fact Questionnaire-2 (HDFQ-2) is a 25-item measure contains true/false questions that were developed to assess participants' knowledge of major risk factors for the development of CHD. Each true/false question that was correctly answered was scored as 4 points, for a maximum possible score of 100, indicting a higher level of knowledge. Any questions that were either unanswered or unsure were scored as incorrect. The HDFQ-2 has demonstrated adequate internal consistency with Cronbach alpha of 0.84 and good test-rested reliability with intraclass correlation coefficient (ICC) of 0.89.
Heart Disease Fact Questionnaire-2 (HDFQ-2) | 6th months from the baseline
  Heart Disease Fact Questionnaire-2 (HDFQ-2) is a 25-item measure contains true/false questions that were developed to assess participants' knowledge of major risk factors for the development of CHD. Each true/false question that was correctly answered was scored as 4 points, for a maximum possible score of 100, indicting a higher level of knowledge. Any questions that were either unanswered or unsure were scored as incorrect. The HDFQ-2 has demonstrated adequate internal consistency with Cronbach alpha of 0.84 and good test-rested reliability with intraclass correlation coefficient (ICC) of 0.89.
Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire | baseline
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire was developed to provide a way to track cardiovascular risk factors. It contains 20 questions to assess participants' heart-related lifestyle status including exercise, cholesterol, tobacco use, alcohol consumption, and exercise activity. Findings form a recent systematic literature review of published articles from 2004 to 2011 detailing the test of reliability and validity of BRFSS indicated that the questionnaire has good reliability and validity.
Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire | 4th week from the baseline
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire was developed to provide a way to track cardiovascular risk factors. It contains 20 questions to assess participants' heart-related lifestyle status including exercise, cholesterol, tobacco use, alcohol consumption, and exercise activity. Findings form a recent systematic literature review of published articles from 2004 to 2011 detailing the test of reliability and validity of BRFSS indicated that the questionnaire has good reliability and validity.
Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire | 6th months from the baseline
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire was developed to provide a way to track cardiovascular risk factors. It contains 20 questions to assess participants' heart-related lifestyle status including exercise, cholesterol, tobacco use, alcohol consumption, and exercise activity. Findings form a recent systematic literature review of published articles from 2004 to 2011 detailing the test of reliability and validity of BRFSS indicated that the questionnaire has good reliability and validity.
Perceived Stress Scale-10 item (PSS-10) | baseline
  Perceived Stress Scale (PSS-10) is the most widely used instrument for measuring an individual's perception of the stress. The PSS consists of 10 items using a 5-point Liker scale with the higher the score indicating higher level of stress. It has been translated into different languages and the reliability and validity of the scale have been well established with Cronbach alpha greater than 0.80 being reported by majority of the studies.
Perceived Stress Scale-10 item (PSS-10) | 4th week from the baseline
  Perceived Stress Scale (PSS-10) is the most widely used instrument for measuring an individual's perception of the stress. The PSS consists of 10 items using a 5-point Liker scale with the higher the score indicating higher level of stress. It has been translated into different languages and the reliability and validity of the scale have been well established with Cronbach alpha greater than 0.80 being reported by majority of the studies.
Perceived Stress Scale-10 item (PSS-10) | 6th months from the baseline
  Perceived Stress Scale (PSS-10) is the most widely used instrument for measuring an individual's perception of the stress. The PSS consists of 10 items using a 5-point Liker scale with the higher the score indicating higher level of stress. It has been translated into different languages and the reliability and validity of the scale have been well established with Cronbach alpha greater than 0.80 being reported by majority of the studies.

OTHER OUTCOMES:
Age | Baseline
  Age
Gender | Baseline
  Gender
Marital Status | Baseline
  Marital status
Occupation | Baseline
  Occupation
Ethinicity | Baseline
  Ethnicity
Monthly income | Baseline
  Monthly income in Singapore dollars
Education level | Baseline
  Highest educational level
BMI | Baseline
  BMI in kg/m^2
Feedback about the Care4Heart app | 6th months from the baseline
  A short questionnaire will be used to obtain feedback about the user experience and overall evaluation of the app from participants at 6-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Wenru Wang, PhD, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreou E, Alexopoulos EC, Lionis C, Varvogli L, Gnardellis C, Chrousos GP, Darviri C. Perceived Stress Scale: reliability and validity study in Greece. Int J Environ Res Public Health. 2011 Aug;8(8):3287-98. doi: 10.3390/ijerph8083287. Epub 2011 Aug 11. PMID 21909307
- [Background] Awad A, Al-Nafisi H. Public knowledge of cardiovascular disease and its risk factors in Kuwait: a cross-sectional survey. BMC Public Health. 2014 Nov 4;14:1131. doi: 10.1186/1471-2458-14-1131. PMID 25367768
- [Background] Beatty AL, Fukuoka Y, Whooley MA. Using mobile technology for cardiac rehabilitation: a review and framework for development and evaluation. J Am Heart Assoc. 2013 Nov 1;2(6):e000568. doi: 10.1161/JAHA.113.000568. No abstract available. PMID 24185949
- [Background] Bunker SJ, Colquhoun DM, Esler MD, Hickie IB, Hunt D, Jelinek VM, Oldenburg BF, Peach HG, Ruth D, Tennant CC, Tonkin AM. "Stress" and coronary heart disease: psychosocial risk factors. Med J Aust. 2003 Mar 17;178(6):272-6. doi: 10.5694/j.1326-5377.2003.tb05193.x. PMID 12633484
- [Background] Chomutare T, Fernandez-Luque L, Arsand E, Hartvigsen G. Features of mobile diabetes applications: review of the literature and analysis of current applications compared against evidence-based guidelines. J Med Internet Res. 2011 Sep 22;13(3):e65. doi: 10.2196/jmir.1874. PMID 21979293
- [Background] Chyun D, Lacey KO, Katten DM, Talley S, Price WJ, Davey JA, Melkus GD. Glucose and cardiac risk factor control in individuals with type 2 diabetes: implications for patients and providers. Diabetes Educ. 2006 Nov-Dec;32(6):925-39. doi: 10.1177/0145721706295016. PMID 17102160
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Fleg JL, Forman DE, Berra K, Bittner V, Blumenthal JA, Chen MA, Cheng S, Kitzman DW, Maurer MS, Rich MW, Shen WK, Williams MA, Zieman SJ; American Heart Association Committees on Older Populations and Exercise Cardiac Rehabilitation and Prevention of the Council on Clinical Cardiology, Council on Cardiovascular and Stroke Nursing, Council on Lifestyle and Cardiometabolic He. Secondary prevention of atherosclerotic cardiovascular disease in older adults: a scientific statement from the American Heart Association. Circulation. 2013 Nov 26;128(22):2422-46. doi: 10.1161/01.cir.0000436752.99896.22. Epub 2013 Oct 28. No abstract available. PMID 24166575
- [Background] Gough D. (2011). Coronary heart disease. Practice Nurse 41(1), 12-17
- [Background] Ghanem F.A., & Movahed A. (2009). Prevention of Coronary Heart Disease. In Movahed, A., Gnanasegaran, G., Buscombe, J., & Hall, M. Integrating Cardiology for Nuclear Medicine Physicians. Springer Berlin Heidelberg. P. 419-423.
- [Background] Centres of Disease Control and Prevention (2013). Behavioural Risk Factors Surveillance System Questionnaire. Retrieved from http://www.cdc.gov/brfss. Oct. 2013.
- [Background] Ministry of Health (2014). Health Matters. Retrieved from ttp://mohsingapore.sg/2012/02/living-healthily/ January. 2014.
- [Background] Infocomm Development Authority of Singapore (2013). iN2015 Masterplan. Retrieved from: http://www.ida.gov.sg/Infocomm-Landscape/iN2015-Masterplan on 01 February 2014.
- [Background] Ministry of Health Singapore (2014). Principal Causes of Death 2013; Available from: http://www.moh.gov.sg/content/moh_web/home/statistics/Health_Facts_Singapore/Principal_Causes_of_Death.html.
- [Background] Polit D. F., & Beck C. T (2014). Essentials of Nursing Research: Methods, Appraisal, and Utilization. 8th edn. Philadelphia: Lippincott.
- [Background] Peck AD. One-touch access to a world of resources: mobile health apps streamline workflows. Med Econ. 2011 Sep 10;88(17):S7-8, S10-1. No abstract available. PMID 22053522
- [Background] Pierannunzi C, Hu SS, Balluz L. A systematic review of publications assessing reliability and validity of the Behavioral Risk Factor Surveillance System (BRFSS), 2004-2011. BMC Med Res Methodol. 2013 Mar 24;13:49. doi: 10.1186/1471-2288-13-49. PMID 23522349
- [Background] Rosenstock IM, Strecher VJ, Becker MH. Social learning theory and the Health Belief Model. Health Educ Q. 1988 Summer;15(2):175-83. doi: 10.1177/109019818801500203. PMID 3378902
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Singapore Heart Foundation (2011). Deaths from Cardiovascular Disease. Retrieved from http://www.myheart.org.sg/heart-facts/statistics/ Oct. 2011.
- [Background] Singapore Heart Foundation (2014). Heart4Life Phase 1. Retrieved from http://www.myheart.org.sg/article/heart-safe-singapore/heart4life-mobile-app/about/186/ January 2014.
- [Background] Smeltzer S. C., Bare B. G., Hinkle J. L., & Cheever K. H. (2010). Brunner & Suddarth's textbook of medical surgical nursing 12th edn. Wallnut Street, Philadelphia: PA.
- [Background] Wagner J, Lacey K, Chyun D, Abbott G. Development of a questionnaire to measure heart disease risk knowledge in people with diabetes: the Heart Disease Fact Questionnaire. Patient Educ Couns. 2005 Jul;58(1):82-7. doi: 10.1016/j.pec.2004.07.004. PMID 15950840
- [Background] World Health Organization (2014). The top 10 causes of death. (Fact sheet No. 310). Retrieved from: http://www.who.int/mediacentre/factsheets/fs310/en/